CLINICAL TRIAL: NCT04558736
Title: Haploidentical Donor Hematopoietic Cell Transplantation for Patients With Severe Aplastic Anemia
Brief Title: Haploidentical HCT for Severe Aplastic Anemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HAPSAA
Record Dates: First submitted 2020-09-09; First posted 2020-09-22 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Aplastic Anemia; Bone Marrow Failure Syndrome
Keywords: Haploidentical Transplant
MeSH Terms: conditions — Anemia, Aplastic; Bone Marrow Failure Disorders | interventions — Antilymphocyte Serum; thymoglobulin; fludarabine; Cyclophosphamide; Mesna; Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Haploidentical HCT (Experimental): To assess the safety and efficacy of haploidentical donor transplantation for patients with severe aplastic anemia who lack an available HLA-matched donor. The goal of this study is to develop a novel, reduced-toxicity, post-transplant pharmacologic immunosuppression (GVHD prophylaxis)- free, highly tolerogenic haploidentical transplant regimen that is associated with few post- transplant complications or late toxicities and is available promptly to all patients, irrespective of matched donor availability.
  Cells for infusion are prepared using the CliniMACS System.
  Interventions: Drug: Anti-Thymocyte Globulin (Rabbit); Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Mesna; Drug: G-CSF; Radiation: Total Lymphoid Irradiation (TLI); Device: CliniMACS; Biological: HPC, A Infusion; Biological: CD45RA-depleted DLI

INTERVENTIONS:
Drug: Anti-Thymocyte Globulin (Rabbit) — Given intravenously (IV)
  Other Names: thymoglobulin; rabbit ATG
Drug: Fludarabine — Given intravenously (IV)
  Other Names: Fludara Flu Dara
Drug: Cyclophosphamide — Given intravenously (IV)
  Other Names: CYTOXAN
Drug: Mesna — Given intravenously (IV)
  Other Names: MESNEX
Drug: G-CSF — Filgrastim is a human granulocyte colony-stimulating factor (G-CSF), produced by recombinant DNA technology. Dosage and Route of Administration: 5mcg/kg subcutaneous or intravenous daily until ANC >2000 for 2 consecutive days, or as clinically indicated
  Other Names: Neupogen; Filgrastim
Radiation: Total Lymphoid Irradiation (TLI) — TLI will be given at 800 cGy total dose in 4 fractions.
  Other Names: TLI
Device: CliniMACS — The mechanism of action of the CliniMACS Cell Selection System is based on magnetic-activated cell sorting (MACS). The CliniMACS device is a powerful tool for the isolation of many cell types from heterogeneous cell mixtures, (e.g. apheresis products). These can then be separated in a magnetic field using an immunomagnetic label specific for the cell type of interest, such as CD3+ human T cells.
  Other Names: Cell Selection System
Biological: HPC, A Infusion — Given intravenously Day 0-HPC, A Infusion (TCR αβ+/CD19+-depleted graft)
Biological: CD45RA-depleted DLI — CD45RA-depleted DLI will be given at least ONE week after engraftment

SUMMARY:
This study is a prospective, single center phase II clinical trial in which patients with Severe Aplastic Anemia (SAA) ) will receive a haploidentical transplantation. The purpose of this study is to learn more about newer methods of transplanting blood forming cells donated by a family member that is not fully matched to the patient. This includes studying the effects of the chemotherapy, radiation, the transplanted cell product and additional white blood cell (lymphocyte) infusions on the patient's body, disease and overall survival. The primary objective is to assess the rate of engraftment at 30 days and overall survival (OS) and event free survival (EFS) at 1 year post-hematopoietic cell transplantation (HCT).

Primary Objectives

* To estimate the rate of engraftment at 30 days after TCR αβ+ T-cell-depleted graft infusion in patients receiving a single dose of post graft infusion cyclophosphamide.
* To estimate the overall survival and event free survival at 1-year post transplantation.

Secondary Objectives

* To calculate the incidence of acute and chronic GVHD after HCT.
* To calculate the rate of secondary graft rejection at 1-year post transplantation
* To calculate the cumulative incidence of viral reactivation (CMV, EBV and adenovirus).
* To describe the immune reconstitution after TCR αβ+ T-cell-depleted graft infusion at 1 month, 3 months, 6 months, 9 months, and 1 year.

Exploratory Objectives

* To longitudinally assess the phenotype and epigenetic profile of T-cells in SAA patients receiving HCT for SAA.
* To assess the phenotype and epigenetic profile of T-cells in DLI administered to SAA patients post HCT.
* To longitudinally assess CD8 T cell differentiation status in SAA patients using an epigenetic atlas of human CD8 T cell differentiation.
* To examine the effector functions and proliferative capacity of CD8 T cells isolated from SAA patients before and after DLI.
* Quantify donor derived Treg cells at different time points in patients received HCT.
* Determine Treg activation status at different stages after HCT.
* Are specific features of the DLI product associated with particular immune repertoire profiles post-transplant?
* How does the diversity and functional profile of the DLI product alter the response to pathogens in the recipient?
* Do baseline features of the recipient's innate and adaptive immune cells correlate with post-transplant immune repertoires and response profiles?

DETAILED DESCRIPTION:
Immunosuppressant therapy (IST) is the main treatment for SAA for patients who do not have an HLA-matched sibling donor available for transplant. But some patients with SAA do not respond to IST and some others relapse after IST. HCT using an unrelated but HLA-matched donor is the only curative option for these patients but many patients lack a suitable HLA-matched donor. St Jude is trying to increase donor options for these patients by using novel therapeutic strategies by combining two widely used of GVHD prophylaxis methods: i) selective T cell depletion and ii) use of post-transplant cyclophosphamide. This will allow expansion of the donor pool to include haploidentical donors as well as reduce the risk of GVHD. The goal of this protocol is to test whether combining these GVHD prophylaxis approaches will allow use of haploidentical donors, reduce risk of GVHD, reduce transfusion dependence and improve immune reconstitution.

For this study chemotherapy, antibodies and radiation will be given to prepare the body to receive donor cells. Participants will then be given the donor cell infusion.

Patients will receive two types of donor blood cell products - a progenitor blood cell infusion and then a donor lymphocyte infusion. Both the progenitor blood cell and the donor lymphocyte infusion will be processed in a laboratory at St. Jude using a machine called the CliniMACS™.

In this clinical trial, participants will receive a special type of progenitor blood cells (called TCRαβ- depleted blood cells) from the donor.

After the donor progenitor cells have started to grow within the body (engraftment), participants will receive a second product that contains mature immune cells. These immune cells called CD45RA-depleted lymphocytes or donor lymphocyte infusion (DLI) will help fight infections in the body after the transplant and strengthen the developing immune system.

ELIGIBILITY:
Inclusion Criteria for Transplant Recipient

1. Age less than or equal to 21 years at time of enrollment.
2. Confirmed diagnosis of SAA or a single lineage cytopenia

   (a) SAA or single lineage cytopenia will be defined as follows:
   * i. Bone marrow cellularity < 25% or hypocellular marrow for age, AND
   * ii. One or more of the following (in peripheral blood): (i) Neutrophils < 0.5 x10^9/L (ii) Platelets < 20 x10^9/L, or platelet transfusion dependence (iii) Hemoglobin <8g/dL, or red blood cell transfusion dependence
3. Does not have a suitable HLA-matched sibling donor (MSD) or volunteer 10/10 HLA-matched unrelated donor (MUD) available in the necessary time for progenitor cell donation.
4. Failed at least one trial of immunosuppressive therapy (IST) by being refractory (persistence of severe cytopenias and fulfillment of SAA disease criteria at least 3 months after initial IST) or having relapsed (initial improvement of cytopenias after first-line IST but then a later return to fulfillment of SAA disease criteria when IST is decreased or ceased). IST could have included ATG based regimens, calcineurin inhibitors and/or other higher dose therapy directed at the treatment of primary SAA. Patients with very severe aplastic anemia who are likely not to benefit from IST do not need to have failed a trial of IST and can proceed directly to HCT if they meet the rest of the criteria.
5. Has a suitable single haplotype matched (≥ 3 of 6) family member donor.
6. Patient and/or legal guardian must sign informed consent for HCT.
7. Adequate organ function defined as:

   1. Left ventricular ejection fraction > 40% or shortening fraction ≥ 25%.
   2. Creatinine clearance (CrCl) or glomerular filtration rate (GFR) ≥ 50 ml/ min/1.73m2.
   3. Forced vital capacity (FVC) ≥ 50% of predicted value; or pulse oximetry
   4. ≥ 92% on room air if patient is unable to perform pulmonary function testing.
   5. Karnofsky or Lansky (age-dependent) performance score ≥ 50.
   6. Bilirubin ≤ 3 times the upper limit of normal for age.
   7. Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) ≤ 5 times the upper limit of normal for age.
8. Females and males of childbearing potential must agree to practice 2 effective methods of contraception at the same time or agree to abstinence until after the last dose of chemotherapy has been administered

Exclusion Criteria for Transplant Recipient:

1. Diagnosis of Fanconi anemia. Fanconi anemia must be excluded by diepoxybutane (DEB) or equivalent testing.
2. Known clinical or genetic diagnosis of dyskeratosis congenita
3. Clonal cytogenetic abnormalities consistent with pre-myelodysplastic syndrome (pre- MDS) or MDS on marrow examination (e.g. Monosomy 7).
4. Diagnosis of myelodysplastic syndrome (MDS).
5. Presence of anti-donor HLA antibodies (positive anti-donor HLA antibody is defined as a positive cross-match test of any titer by complement- dependent cytotoxicity or flow cytometric testing or the presence of anti- donor HLA antibody to the high expression loci HLA-A, B, C, DRB1, or DPB1 with mean fluorescence intensity (MFI) > 1000 by solid phase immunoassay).
6. Prior allogeneic hematopoietic cell transplant.
7. Prior solid organ transplant.
8. Known life-threatening reaction (i.e., anaphylaxis) to ATG that would prohibit use for the patient.
9. Uncontrolled bacterial, viral, or fungal infection at the time of enrollment. Uncontrolled is defined as progression or no clinical improvement on appropriate medical treatment.
10. Female patients who are pregnant (per institutional practice) or breast- feeding.
11. Prior malignancies except resected basal cell carcinoma or treated cervical carcinoma in situ. Cancer treated with curative intent > 5 years previously will be allowed. Cancer treated with curative intent ≤ 5 years previously will not be allowed unless approved by the PI.
12. Alemtuzumab or ATG within 2 weeks of enrollment.

Inclusion Criteria for Haploidentical Donor

1. At least single haplotype matched (≥ 3 of 6) family member.
2. At least 18 years of age.
3. HIV negative.
4. Not pregnant as confirmed by negative serum or urine pregnancy test within 14 days prior to enrollment (if female).
5. Not breast feeding.
6. Related donors must be ruled out for telomere disease by appropriate clinical and diagnostic measures (for example, clinical evaluation, telomere length testing, genetic testing, and/or bone marrow examination).
7. The HAPLO donor and/or legal guardian must be able to sign informed consent documents.
8. The potential HAPLO donor must be willing and able to donate PBSCs.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Estimated)
Dates: Start 2021-01-21 (Actual); Primary Completion 2029-07-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
Engraftment | 30 days
  Rate of patients engrafting at day 30 after TCR αβ+ T-cell-depleted graft infusion in patients receiving a single dose of post graft infusion cyclophosphamide.
Overall and event free survival | 1 year
  Rate of overall survival and event free survival at 1-year post transplantation.

SECONDARY OUTCOMES:
Graft vs host disease | 1 year
  Incidence of acute and chronic GVHD after hematopoietic cell transplant
Graft rejection | 1 year
  Rate of secondary graft rejection at 1-year post transplantation
Viral reactivation | 1 year
  Cumulative incidence of viral reactivation post-transplant (CMV, EBV and adenovirus)
Immune reconstitution | 1 year
  We will record immune reconstitution parameters, including the order and magnitude of recovery of the different subtypes of leukocytes. Results will be summarized by descriptive statistics. The pattern of immune reconstitution will be evaluated using longitudinal approaches such as mixed effect models or generalized estimating equation (GEE) approach.

CONTACTS AND LOCATIONS:
Overall Officials: Amr Qudeimat, MD, Principal Investigator — St. Jude Children's Research Hospital; Akshay Sharma, MBBS, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols